CLINICAL TRIAL: NCT02777008
Title: A Two-Part Single Center, Randomized, Sequential, Single and Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of CTP-543 in Healthy Volunteers
Brief Title: Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of CTP-543 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Concert Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CP543.1001
Record Dates: First submitted 2016-05-16; First posted 2016-05-19 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CTP-543 Single Dose (Experimental): Single oral dose
  Interventions: Drug: CTP-543; Drug: Placebo for CTP-543
- CTP-543 Multiple Dose (Experimental): Multiple oral dose for 7 consecutive days
  Interventions: Drug: CTP-543; Drug: Placebo for CTP-543

INTERVENTIONS:
Drug: CTP-543
Drug: Placebo for CTP-543

SUMMARY:
Single- and multiple-ascending dose study of CTP-543 in healthy volunteers.

DETAILED DESCRIPTION:
This two-part study will assess, in healthy volunteers, under fasted conditions, and in a sequential manner, the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of single- and multiple-ascending doses of CTP-543.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males and females between 18 and 50 years of age, inclusive
* Body weight ≥ 50 kg and BMI within the range of 18 to 30 kg/m2, inclusive

Exclusion Criteria:

* History of clinically significant central nervous system (eg, seizures), cardiac, pulmonary, metabolic, renal, hepatic, or gastrointestinal (GI) conditions
* PR interval > 220 msec or QRS duration > 120 msec or QTcF interval > 450 msec obtained at screening visit or prior to the first dose of study drug
* History of herpes zoster
* Hemoglobin, white blood cell, or platelet levels below the lower reference limit at screening or prior to the first dose of study drug
* Liver function tests greater than the upper limit of normal
* Positive blood screen for human immunodeficiency virus (HIV antibody), hepatitis B virus surface antigen, or hepatitis C virus antibody
* Urinalysis positive for protein or glucose
* A positive screen for alcohol, drugs of abuse, or tobacco use
* Donation of blood, plasma or other blood products prior to screening
* A positive tuberculosis test

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2016-05; Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 24 hours
Measurement of CTP-543 exposure in plasma under fasted conditions | 24 hours

OTHER OUTCOMES:
The relationship between CTP-543 drug concentration and effect | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Hamilton, Study Director — Concert Pharmaceuticals, Inc.
Locations (1):
- Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No